CLINICAL TRIAL: NCT07111416
Title: Personalizing A1c Using Hematologic Indices and CGM for Accurate Diabetes Diagnosis (PRECISE DM Dx)
Brief Title: Personalizing A1c Using Hematologic Indices and CGM for Accurate Diabetes Diagnosis
Acronym: PRECISE DM DX
Status: Not yet recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Abbott Diabetes Care (Industry)
Responsible Party: Principal Investigator, Marie McDonnell, Associate Professor, Brigham and Women's Hospital
Other Study IDs: 2025P001596
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

SUMMARY:
The goal of this observational study is to learn why some adults over the age of 65, have A1c tests that do not match up with their blood glucose levels, also known as 'A1c-glucose discordance'.

The main question it aims to answer is:

Could alternative tests like CGM or personalized A1c provide more accurate diabetes screening in this population?

Participants will be asked to perform blood tests every week to two weeks and wear a CGM for up to 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years of age or older
* A1c 5.3% - 7.4% without a diagnosis on the problem list and/or current or prior treatment for diabetes
* Evidence of A1c discordance by meeting one of two criteria developed by an EHR based algorithm
* At least five (5) HbA1c values and three (3) CBC values available in the EHR in the previous 10 years
* Willingness to wear an Abbott Freestyle Libre 3 System Sensor for up to 48 days
* Willingness to consent to data collection using the electronic health record and sign a medical release to obtain future medical records from other health care facilities

Exclusion Criteria:

* Known or suspected diabetes of other causes (type 1 diabetes, pancreatogenic diabetes, monogenic diabetes, etc.)
* Clinically significant anemia based on most recent hematocrit (M = <38%, F <33%) and/or hemoglobin (M = <12 g/dL, F = <10 g/dL) within the last 12 months
* Condition with short life expectancy
* Blood (hematologic) malignancy
* rtCGM-interference agents per manufacturer (e.g., high dose vitamin C)
* Unstable psychiatric or medical condition
* Active treatment for cancer, planned treatment for cancer, or recent active cancer with a likelihood of recurrence or progression, that, in the opinion of the site investigator, would interfere with study therapy prior to 2029

  * Allowed Exceptions: Treated cancer with no evidence of disease, no evidence of disease progression, and no planned change in therapy. Examples of allowable cancers include:

    * Breast cancer stable after active treatment, managed with long-term anti-estrogen therapy
    * Prostate cancer being observed
    * Stage 0 or 1 tumors status post resection or other definitive treatment
    * Other similarly stable cancer comorbidities

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Individuals 65 years of age and older, who have evidence of A1c-glucose discordance without either a diagnosis of type 2 diabetes or current/ prior treatment for type 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Calculate the Mean Absolute Difference Between A1c-Derived Estimated Average Glucose (eAG) and CGM-Derived eAG | From 1 week after enrollment to the end of their enrollment at either week 5 or week 10
  Determine the mean absolute difference between estimated average glucose (eAG) calculated from hemoglobin A1c and eAG derived from Continuous Glucose Monitoring (CGM) data. This measure will be assessed among participants suspected of having discordance between A1c values and actual blood glucose levels.